CLINICAL TRIAL: NCT03322657
Title: Sugammadex Versus Neostigmine for Reversal of Rocuronium Neuromuscular Block in Patients Having Catheter-based Neurointerventional Procedures
Brief Title: Sugammadex Versus Neostigmine for Reversal of Rocuronium Neuromuscular
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Ehab Farag, MD, Ehab Farag, M.D., The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 17-764
Record Dates: First submitted 2017-10-13; First posted 2017-10-26 (Actual); Results first posted 2021-04-08 (Actual); Last update posted 2021-11-16 (Actual); Status verified 2021-10

CONDITIONS: Neuromuscular Blockade; Anesthesia
Keywords: Sugammadex; Neostigmine; Reversal of neuromuscular block
MeSH Terms: interventions — Neostigmine; Glycopyrrolate; Sugammadex

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Neostigmine with glycopyrrolate (Active Comparator): Neostigmine 0. 07 mg/kg with glycopyrrolate 0.01 mg/kg with ceiling dose of 5 mg neostigmine with 1 mg of glycopyrrolate at the end surgery
  Interventions: Drug: Neostigmine; Drug: Glycopyrrolate
- Sugammadex (Experimental): Sugammadex 4 mg/kg at the end surgery
  Interventions: Drug: Sugammadex

INTERVENTIONS:
Drug: Neostigmine — Neostigmine injection
  Arms: Neostigmine with glycopyrrolate
Drug: Glycopyrrolate — Glycopyrrolate injection
  Arms: Neostigmine with glycopyrrolate
Drug: Sugammadex — Sugammadex injection
  Arms: Sugammadex

SUMMARY:
The aim of this study is to evaluate whether the use of Sugammadex for reversing the neuromuscular blocking effects of rocuronium during neurointerventional procedures can speed recovery of neuromuscular function. Half of participates will receive Neostigmine with glycopyrrolate, while the other half will receive Sugammadex.

DETAILED DESCRIPTION:
Incomplete recovery from neuromuscular blocking agents (NMBAs) residual block after anesthesia and surgery continues to be a common problem in the postanesthesia care (PACU).

Neostigmine remains the most common acetylcholinesterase inhibitor in the United States. However, administration of the drug significantly impairs genioglossus muscle activity when administered after full recovery from neuromuscular block. Moreover, doses of neostigmine exceeding 0.06 mg/kg increase the risk of respiratory complications independent of NMBAs effects.

Sugammadex is a modified γ-cyclodextrin that rapidly reverses that effect of the steroidal nondepolarizing NMBAs rocuronium and vecuronium. Sugammadex forms a stable, inactive 1:1 complex with rocuronium or vecuronium, reducing the amount of free NMBA available to bind to nicotinic acetylcholine receptors at the neuromuscular junction. Unlike neostigmine, sugammadex completely reverses even dense neuromuscular blocks.

Patients having catheter-based neurointerventional procedures are kept deeply anesthetized. It is common to find patients nearly completely paralyzed at the end of neurointerventional procedures and have a markedly delayed emergence while waiting for muscle function to recover sufficiently to safely antagonize with neostigmine.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years;
* American Society of Anesthesiologists (ASA) physical status 1-3;
* Scheduled for catheter-based neurointerventional procedures including coiling and stent insertion;
* General anesthesia.

Exclusion Criteria:

* Suspected difficult intubation;
* Neuromuscular disorder;
* Renal impairment creatinine ≥ 2 mg /dl;
* Hepatic dysfunction;
* History of malignant hyperthermia;
* Allergy to neuromuscular blocking drugs, Sugammadex, neostigmine or glycopyrrolate;
* Perioperative respiratory infections and/or pneumonia;
* Intubated or unresponsive;
* Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2017-11-14 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Farag E, Rivas E, Bravo M, Hussain S, Argalious M, Khanna S, Seif J, Pu X, Mao G, Bain M, Elgabaly M, Esa WAS, Sessler DI. Sugammadex Versus Neostigmine for Reversal of Rocuronium Neuromuscular Block in Patients Having Catheter-Based Neurointerventional Procedures: A Randomized Trial. Anesth Analg. 2021 Jun 1;132(6):1666-1676. doi: 10.1213/ANE.0000000000005533. PMID 34032663

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Neostigmine With Glycopyrrolate | Sugammadex
Started | 34 | 35
Completed | 33 | 35
Not Completed | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neostigmine With Glycopyrrolate | Sugammadex | Total
Number analyzed (Participants) | 33 | 35 | 68
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (12) | 54 (15) | 56 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 27 | 46
  Male | 14 | 8 | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Afirican American | 3 | 3 | 6
  Race: Asian | 1 | 0 | 1
  Race: Caucasian | 29 | 32 | 61
Weight [Mean (Standard Deviation); unit: kg] | 90 (32) | 92 (38) | 91 (35)
ASA [Count of Participants; unit: Participants] — American Society of Anesthesiologists physical status is to assess and communicate a patient's pre-anesthesia medical co-morbidities. This status has a grade from I to VI, where I mean a normal healthy patient and VI means a declared brain-dead patient whose organs are being removed for donor purposes.
  Participants
    II | 3 | 3 | 6
    III | 32 | 32 | 64
Arterial hypertension [Count of Participants; unit: Participants] | 20 | 23 | 43
Asthma [Count of Participants; unit: Participants] | 3 | 3 | 6
Chronic pulmonary disease [Count of Participants; unit: Participants] | 5 | 3 | 8
Obstructive sleep apnea [Count of Participants; unit: Participants] | 6 | 4 | 10
Diabetes mellitus [Count of Participants; unit: Participants] | 4 | 6 | 10
Myocardial infarction [Count of Participants; unit: Participants] | 1 | 1 | 2
Ischemic heart disease [Count of Participants; unit: Participants] | 0 | 2 | 2
Neurologic diseases [Count of Participants; unit: Participants] | 9 | 7 | 16
Chronic pain requiring opioids [Count of Participants; unit: Participants] | 0 | 1 | 1
Current smoker [Count of Participants; unit: Participants] | 5 | 8 | 13
Current recreational drug user [Count of Participants; unit: Participants] | 0 | 0 | 0
Alcohol abuse [Count of Participants; unit: Participants] | 0 | 1 | 1
Cancer [Count of Participants; unit: Participants] | 0 | 2 | 2
No medical history [Count of Participants; unit: Participants] | 3 | 3 | 6
Intraoperative remifentanil [Count of Participants; unit: Participants] — Intraoperative remifentanil use could be related to our outcome and it was before the treatment, thus we think it was important to report it as baseline measures.
  Participants | 14 | 8 | 22
Intraoperative remifentanil, μg [Median (Inter-Quartile Range); unit: μg] — Intraoperative remifentanil use could be related to our outcome and it was before the treatment, thus we think it was important to report it as baseline measures.
  μg | 0 [0 to 542] | 0 [0 to 0] | 0 [0 to 444]
Intraoperative fentanyl [Count of Participants; unit: Participants] — Intraoperative fentanyl use could be related to our outcome and it was before the treatment, thus we think it was important to report it as baseline measures.
  Participants | 33 | 35 | 68
Intraoperative fentanyl, mg [Median (Inter-Quartile Range); unit: mg] — Intraoperative fentanyl use could be related to our outcome and it was before the treatment, thus we think it was important to report it as baseline measures.
  mg | 0.10 [0.07 to 0.12] | 0.10 [0.09 to 0.15] | 0.10 [0.08 to 0.15]
Intraoperative propofol, mg [Median (Inter-Quartile Range); unit: mg] — Intraoperative propofol use could be related to our outcome and it was before the treatment, thus we think it was important to report it as baseline measures.
  mg | 200 [150 to 230] | 200 [150 to 242] | 200 [150 to 241]
Intraoperative midazolam, mg [Median (Inter-Quartile Range); unit: mg] — Intraoperative midazolam use could be related to our outcome and it was before the treatment, thus we think it was important to report it as baseline measures.
  mg | 0 [0 to 1] | 0 [0 to 2] | 0 [0 to 2]
Intraoperative Phenylephrine [Count of Participants; unit: Participants] — Intraoperative phenylephrine use could be related to our outcome and it was before the treatment, thus we think it was important to report it as baseline measures.
  Participants | 25 | 25 | 50
Intraoperative Ephedrine [Count of Participants; unit: Participants] — Intraoperative ephedrine use could be related to our outcome and it was before the treatment, thus we think it was important to report it as baseline measures.
  Participants | 7 | 9 | 16
Intraoperative Norepinephrine [Count of Participants; unit: Participants] — Intraoperative norepinephrine use could be related to our outcome and it was before the treatment, thus we think it was important to report it as baseline measures.
  Participants | 0 | 0 | 0
Time-weighted average minimum alveolar concentration [Median (Inter-Quartile Range); unit: percent at 1 atmosphere] — time-weighted average minimum alveolar concentration could be related to our outcome and it was before the treatment, thus we think it was important to report it as baseline measures.
  percent at 1 atmosphere | 0.79 [0.68 to 0.88] | 0.78 [0.69 to 0.87] | 0.78 [0.69 to 0.88]

OUTCOME MEASURES:

1. Primary Outcome: Time in Minutes to Reach Train of Four (TOF) Ratio ≥ 0.9 After the Administration of Reversal Agent
Description: The primary outcome was a time-to-TOF ratio ≥ 0.9 after the administration of the reversal agent. The TOF ratio was measured in a continuous manner every 12 seconds from the administration of the reversal drug until TOF ratio ≥ 0.9 or until 90 minutes after administration of the reversal agent.
Time Frame: within 90 minutes after endotracheal extubation
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Neostigmine With Glycopyrrolate | Sugammadex
Number analyzed (Participants) | 33 | 35
minutes | 8 [6 to 10] | 3 [2 to 3]
Statistical Analysis 1: Comparison: Neostigmine With Glycopyrrolate vs Sugammadex; Test type: Superiority; p < 0.001, Cox proportional hazard model; Hazard Ratio (HR) = 3.8, 95% CI 2-sided [2.2 to 6.5]

2. Primary Outcome: TOF Ratio at 90 Min
Description: TOF (train of four), also known as a peripheral nerve stimulator, is used to assess nerve function in patients receiving neuromuscular blocking agents (paralytic medications). Before giving the medications, the baseline must be measured because this tells how much electrical stimulation the patient needs for nerve stimulation without any paralytic on board.
  Our primary outcome TOF ratio between TOF at 90 minutes after the administration of the reversal agent versus the TOF at baseline tells us how well the treatment is working to reverse the rocuronium Neuromuscular. This is a sensitivity analysis of primary analysis.
Time Frame: at 90 minutes after the administration of the reversal agent
Population: Eight patients were removed due to missing TOF at 90 min or TOF count not larger than 4.
Measure: Median (Inter-Quartile Range); unit: ratio
Arm/Group | Neostigmine With Glycopyrrolate | Sugammadex
Number analyzed (Participants) | 28 | 32
ratio | 1.07 [1 to 1.14] | 1.16 [1.02 to 1.26]
Statistical Analysis 1: Comparison: Neostigmine With Glycopyrrolate vs Sugammadex; Test type: Superiority; p = 0.13, Wilcoxon (Mann-Whitney); Median Difference (Final Values) = 6.3, 95% CI 2-sided [-2.0 to 14]

3. Secondary Outcome: The Time for Extubation After Administration of Reversal Agents
Description: Time from administration of reversal agent to tracheal extubation
Time Frame: Up to 4 hours after administration of reversal agents
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | Neostigmine With Glycopyrrolate | Sugammadex
Number analyzed (Participants) | 33 | 35
minutes | 8 [6 to 10] | 8 [6 to 11]
Statistical Analysis 1: Comparison: Neostigmine With Glycopyrrolate vs Sugammadex; Test type: Superiority; p = 0.30, Cox proportional hazard model; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.43 to 1.34]

4. Secondary Outcome: Change of Diaphragmatic Contractility Speed- Sniff (Breathing From the Nose), cm/s
Description: The change of diaphragmatic contractility speed was defined as baseline minus postoperative diaphragmatic contraction.
Time Frame: from baseline to 90 minutes after the administration of the reversal agent
Population: There were 6 (17%) missing in sugammadex group and 5 (15%) missing in neostigmine group on diaphragmatic function outcomes.
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Neostigmine With Glycopyrrolate | Sugammadex
Number analyzed (Participants) | 28 | 29
cm/s | -0.04 (0.85) | 0.29 (1.13)
Statistical Analysis 1: Comparison: Neostigmine With Glycopyrrolate vs Sugammadex; Test type: Superiority; p = 0.21, t-test, 2 sided; Mean Difference (Final Values) = 0.33, 95% CI 2-sided [-0.35 to 1.00]

5. Secondary Outcome: Change of Diaphragmatic Contractility Speed, Deep Breathing From Mouth, cm/s
Description: The change of diaphragmatic contractility speed was defined as baseline minus postoperative diaphragmatic contraction.
Time Frame: from baseline to 90 minutes after the administration of reversal agent
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: cm/s
Arm/Group | Neostigmine With Glycopyrrolate | Sugammadex
Number analyzed (Participants) | 28 | 29
cm/s | -0.02 (1.43) | 0.80 (1.51)
Statistical Analysis 1: Comparison: Neostigmine With Glycopyrrolate vs Sugammadex; Test type: Superiority; p = 0.04, t-test, 2 sided; Mean Difference (Final Values) = 0.82, 95% CI 2-sided [-0.18 to 1.81]

ADVERSE EVENTS:
Time Frame: Until hospital discharge or 30 days after surgery, which came first
Arm/Group | Neostigmine With Glycopyrrolate | Sugammadex
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/35
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/35
Other Adverse Events (participants affected / at risk) | 0/33 | 0/35

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-04-17): https://cdn.clinicaltrials.gov/large-docs/57/NCT03322657/Prot_SAP_000.pdf